CLINICAL TRIAL: NCT01391793
Title: Corticosteroids for Children With Febrile Urinary Tract Infections
Acronym: STARRS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nader Shaikh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Nader Shaikh, Assistant Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01DK087870 (NIH); R01DK087870 (NIH)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Acute Urinary Tract Infection; Urinary Tract Infection
Keywords: Renal scarring; Dexamethasone; Child; Corticosteroids; Pediatric; Urinary tract infection; Escherichia Coli Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Dexamethasone; Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant dexamethasone (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Twice daily for 3 days
  Other Names: Inactive medicine
  Arms: Placebo
Drug: Dexamethasone — 0.15 mg/kg/dose twice daily for 3 days
  Other Names: Prelone; Orapred; Corticosteroid
  Arms: Adjuvant dexamethasone

SUMMARY:
In this study the investigators will determine whether corticosteroids given at the time of urinary tract infection help prevent permanent damage to the kidneys.

DETAILED DESCRIPTION:
Because host inflammatory response is the final and most important step in the formation of renal scars, the use of anti-inflammatory agents may be the best strategy to reduce renal scarring. In animal studies, the use of corticosteroids has been shown to be effective in preventing post-pyelonephritic scarring. We will conduct a randomized, double-blind, placebo-controlled trial to determine the efficacy of 3 days of daily adjuvant dexamethasone on the incidence of renal scarring 4 to 6 months after a first febrile urinary tract infection (UTI). We hypothesize that the proportion of children with UTI who develop renal scarring will be lower among children who are treated with both dexamethasone and antibiotics as compared with children treated with antibiotics alone.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 months to 6 years
* Pyuria: ≥10 white blood cells per cubic millimeter (WBC/mm3) in an uncentrifuged specimen or ≥5 white blood cells per high power field (WBC/hpf) in a centrifuged specimen or ≥1+ leukocyte esterase (LE) on dipstick
* Fever: documented temperature of at least 101 °F or 38.3°C, measured anywhere on the body either at home or at doctor's office within 24 hours of diagnosis

Exclusion Criteria:

* Other concurrent systemic bacterial infection(s) such as meningitis or pneumonia;
* Planned admission to intensive care unit;
* Known bacteremia;
* Previous protocol defined UTI;
* Known major urinary tract anomalies (severe hydronephrosis, ureterocele, urethral valve, solitary or profoundly small kidney, multicystic dysplastic kidney, neurogenic bladder, pelvic or fused kidney);
* Congenital/acquired immunodeficiency;
* Bag urine collection
* Chronic diseases that could potentially interfere with response to therapy, such as chronic gastrointestinal conditions (i.e. malabsorption, inflammatory bowel disease), liver/kidney failure;
* Allergy to dexamethasone
* Antibiotic use within 7 days of enrollment (except if given in the last 48 hours)
* Systemic use of corticosteroids or other immunomodulating agents within 14 days of enrollment
* History of Kawasaki disease
* Sickle cell disease (not trait)

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 546 (Actual)
Dates: Start 2011-09; Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Shaikh, MD, Principal Investigator — University of Pittsburgh
Locations (6):
- United States (6):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nationwide Children's Hospital in Columbus, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Primary Children's Hospital, Salt Lake City, Utah
  - American Family Children's Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaikh N, Liu H, Kurs-Lasky M, Forster CS. Biomarkers for febrile urinary tract infection in children. Pediatr Nephrol. 2022 Jan;37(1):171-177. doi: 10.1007/s00467-021-05173-x. Epub 2021 Jul 12. PMID 34251495
- [Derived] Shaikh N, Shope TR, Hoberman A, Muniz GB, Bhatnagar S, Nowalk A, Hickey RW, Michaels MG, Kearney D, Rockette HE, Charron M, Lim R, Majd M, Shalaby-Rana E, Kurs-Lasky M, Cohen DM, Wald ER, Lockhart G, Pohl HG, Martin JM. Corticosteroids to prevent kidney scarring in children with a febrile urinary tract infection: a randomized trial. Pediatr Nephrol. 2020 Nov;35(11):2113-2120. doi: 10.1007/s00467-020-04622-3. Epub 2020 Jun 15. PMID 32556960

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvant Dexamethasone | Placebo
Started (Randomized to the treatment group) | 271 | 275
Had a Positive Urine Culture | 197 | 188
Completed (Had an outcome Dimercaptosuccinic Acid (DMSA) renal scan 5-24 months from enrollment) | 124 | 131
Not Completed | 147 | 144
Not completed — Ineligible | 3 | 0
Not completed — Urine Culture Negative or Indeterminate | 71 | 87
Not completed — No DMSA | 73 | 57

BASELINE CHARACTERISTICS:
Population: 546 children were randomized; 271 to Adjuvant Dexamethasone and 275 to Placebo. 3 of the 271 were found ineligible post randomization & were withdrawn by the PI. 71 & 87 participants in the respective groups had negative/indeterminate cultures. The remaining 197 & 188 participants had positive urine cultures & were the basis for the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjuvant Dexamethasone | Placebo | Total
Number analyzed (Participants) | 197 | 188 | 385
Age, Customized [Count of Participants; unit: Participants]
  1-23 months | 145 | 132 | 277
  24-47 months | 39 | 32 | 71
  48-71 months | 13 | 24 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 171 | 354
  Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 29
  Not Hispanic or Latino | 181 | 175 | 356
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 41 | 28 | 69
  White | 128 | 126 | 254
  More than one race | 17 | 27 | 44
  Unknown or Not Reported | 0 | 1 | 1
Study Site [Count of Participants; unit: Participants] — Participating clinical study sites included: Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania; Nationwide Children's Hospital,Columbus, Ohio; American Family Children's Hospital, Madison, Wisconsin; Children's National Medical Center, Washington, District of Columbia; Hasbro Children's Hospital, Providence, Rhode Island; and Primary Children's Hospital, Salt Lake City, Utah
  Participants
    Children's Hospital of Pittsburgh, Pittsburgh | 185 | 175 | 360
    Nationwide Children's Hospital, Columbus | 7 | 8 | 15
    American Family Children's Hospital, Madison | 1 | 1 | 2
    Children's National Medical Center, D.C. | 1 | 2 | 3
    Hasbro Children's Hospital, Providence | 1 | 1 | 2
    Primary Children's Hospital, Salt Lake City | 2 | 1 | 3
Maternal Education [Count of Participants; unit: Participants]
  Less than high school | 6 | 11 | 17
  High school graduate or equivalent | 116 | 96 | 212
  College graduate | 66 | 76 | 142
  Unknown | 9 | 5 | 14
Type of Health Insurance [Count of Participants; unit: Participants] — Type of health insurance relates to the child's health insurance.
  Participants
    Private | 81 | 97 | 178
    Public | 108 | 86 | 194
    None | 6 | 3 | 9
    Unknown | 2 | 2 | 4
Duration of Fever [Count of Participants; unit: Participants] — Duration of fever was calculated as the absolute difference between the date and time the participant's fever began and the date and time the participant's urine was collected. The duration was categorized as less than (<) 48 hours or greater than or equal to (>=) 48 hours.
  Participants
    < 48 hours | 110 | 96 | 206
    >= 48 hours | 87 | 92 | 179
Ibuprofen Taken in the Past 24 hours [Count of Participants; unit: Participants]
  No | 88 | 83 | 171
  Yes | 109 | 105 | 214
Escherichia Coli Present in Urine Culture [Count of Participants; unit: Participants]
  No | 10 | 12 | 22
  Yes | 187 | 176 | 363

OUTCOME MEASURES:

1. Primary Outcome: The Distribution of Children With Renal Scarring at the Outcome Dimercaptosuccinic Acid (DMSA) Renal Scan
Description: Renal scarring was defined as decreased uptake of tracer with or without loss of contours. Three radiologists independently reviewed for scarring all DMSA scans that were of adequate quality. For a given kidney, the presence or absence of scarring was the diagnosis endorsed by the majority of readers, i.e. 2 of 3. For a given child, if either kidney or both kidneys were diagnosed with scarring by the majority of readers, then the child was determined to have renal scarring.
Time Frame: The outcome DMSA scan was 5-24 months from enrollment. The mean number of months was 6.1.
Population: The analysis was Intent-to-Treat (ITT). The number of participants is equal to the number of children randomized and eligible who had a positive urine culture at enrollment and a DMSA renal scan, of adequate quality, 5-24 months from the time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Dexamethasone | Placebo
Number analyzed (Participants) | 123 | 131
Participants
  With scarring | 12 | 22
  Without scarring | 111 | 109
Statistical Analysis 1: Comparison: Adjuvant Dexamethasone vs Placebo; Null hypothesis: There is no difference between the two treatment arms regarding the proportion of children with renal scarring at the outcome DMSA renal scan; Test type: Superiority; p = 0.16, Regression, Logistic; The p-value is adjusted for the stratification variable, duration of fever, and for age at baseline (<24 months, >=24 months)

2. Primary Outcome: The Distribution of Children With Severe Renal Scarring at the Outcome Dimercaptosuccinic Acid (DMSA) Renal Scan
Description: Renal scarring was defined as decreased uptake of tracer with or without loss of contours. Scarring was assessed semi-quantitatively by dividing the renal cortex into 12 equal segments. Severe scarring was defined as greater than 4 affected renal segments or global atrophy, i.e. diffuse scarring or shrunken kidney. Three radiologists independently reviewed for scarring all DMSA scans that were of adequate quality. For a given kidney, the presence or absence of severe scarring was the diagnosis endorsed by the majority of readers, i.e. 2 of 3. For a given child, if either kidney or both kidneys were diagnosed with severe scarring by the majority of readers, then the child was determined to have severe renal scarring.
Time Frame: The outcome DMSA scan was 5-24 months from enrollment. The mean number of months was 6.1.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized and eligible who had a positive urine culture at enrollment and a DMSA renal scan, of adequate quality, 5-24 months from the time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Dexamethasone | Placebo
Number analyzed (Participants) | 123 | 131
Participants
  With severe scarring | 0 | 3
  Without severe scarring | 123 | 128
Statistical Analysis 1: Comparison: Adjuvant Dexamethasone vs Placebo; Null hypothesis: There is no difference between the two treatment arms regarding the proportion of children with severe renal scarring at the outcome DMSA renal scan; Test type: Superiority; p = 0.25, Test of equality - 2 Poisson parameters; The method used is a conditional test

3. Secondary Outcome: The Mean Proportion of Children With Renal Scarring at the Outcome Dimercaptosuccinic Acid (DMSA) Renal Scan Taken Across the 3 Radiologists
Description: Renal scarring was defined as decreased uptake of tracer with or without loss of contours. Three radiologists independently reviewed for scarring all DMSA scans that were of adequate quality. For each radiologist, for each child, if either kidney or both kidneys were diagnosed with scarring, then the child was determined to have renal scarring. For each radiologist, the proportion of children with scarring in a given treatment group is the number of children diagnosed with scarring divided by the number of children in the treatment group. The mean proportion of children with scarring in a given treatment group is the average proportion taken across the 3 radiologists.
Time Frame: The outcome DMSA scan was 5-24 months from enrollment. The mean number of months was 6.1.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: proportion of participants with scarring
Arm/Group | Adjuvant Dexamethasone | Placebo
Number analyzed (Participants) | 123 | 131
proportion of participants with scarring | 0.127 (0.050) | 0.204 (0.046)
Statistical Analysis 1: Comparison: Adjuvant Dexamethasone vs Placebo; Null hypothesis: There is no difference between the two treatment arms regarding the mean proportion of children with renal scarring at the outcome DMSA scan taken across the 3 radiologists; Test type: Superiority; p = 0.07, Generalized estimating equations; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Parents were called on days 2,3 and 4 to monitor for adverse events (AEs) after administration of study medication. If the child remained febrile by day 4, daily phone calls were made until the child was afebrile. Monthly phone calls monitored for AEs; parents were reminded to call the 24-hour study line with concerns regarding their child's health. Parents were interviewed at interim visits and at the final 6-month study contact to elicit AEs.
Description: Staff reviewed the child's medical record for any medical care visits since their last study contact for any adverse events. If child was seen or had any new symptoms within 2 weeks of taking study product, the symptoms were reported as adverse events. After 2 weeks of taking study product, if a child was seen for fever or urinary symptoms but not diagnosed with a urinary tract infection these symptoms were reported as an adverse event.
Arm/Group | Adjuvant Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/275
Serious Adverse Events (participants affected / at risk) | 9/271 | 9/275
Other Adverse Events (participants affected / at risk) | 68/271 | 52/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Dexamethasone (N=271) | Placebo (N=275)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 2 (2)
Fever unspecified (General disorders) | 1 (1) | 0 (0)
Fussy infant (General disorders) | 1 (1) | 0 (0)
Kawasaki's disease (General disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Retropharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Poor weight gain in infact (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Posterior urethral values (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 2 (2)
Rash; non-specific skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Dexamethasone (N=271) | Placebo (N=275)
Diarrhea (Gastrointestinal disorders) | 19 (20) | 16 (17)
Fever (General disorders) | 28 (30) | 27 (33)
Fussiness (General disorders) | 27 (29) | 9 (9)
Urinary Tract Infection (UTI) symptoms (Renal and urinary disorders) | 10 (11) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT01391793/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT01391793/ICF_001.pdf